CLINICAL TRIAL: NCT01950338
Title: CHANGES IN SPASTICITY, WIDESPREAD PRESSURE PAIN SENSITIVITY, AND BAROPODOMETRY AFTER DRY NEEDLING IN STROKE PATIENTS
Brief Title: Deep Dry Needling for the Management of Post-stroke Spasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, PROFESSOR, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC 52/2012
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dry needling group (Experimental): The experimental group will receive a single session of DDN with disposable stainless steel needles (0.3mm x 50mm) that will be inserted into the skin over taut bands of the gastrocnemius and tibialis anterior muscles.
  Interventions: Other: Dry needling
- Control group (No Intervention): The control group will not receive any intervention.

INTERVENTIONS:
Other: Dry needling — Once the most painful spot is located within a palpable spastic taut band, the overlying skin is cleaned with alcohol. The needle will be inserted, penetrating the skin about 15-20mm, until the first local twitch response is obtained. Once the first local twitch response is obtained, the needle will be moved up and down (4 to 5 mm. vertical motions with no rotation) in the muscle at approximately 1Hz for 25-30 seconds.
  Arms: Dry needling group

SUMMARY:
Stroke is the leading cause of physical disability, particularly due to the presence of spasticity. Different needling techniques, including the use of Botulinum Toxin A are proposed for the management of spasticity. The presence of spasticity in the lower extremity implies several impairments for standing and walking inducing high disability. No study has investigated the effects of deep dry needling inserted into the targeted spastic musculature in patients with stroke. The investigators will conduct a randomized controlled trial investigating the effects of a single session of deep dry needling over the musculature of the leg on spasticity, widespread pressure pain sensitivity and plantar pressures (baropodometry) in individuals with chronic stroke. The investigators hypothesize that patients receiving a single session of dry needling would exhibit a greater reduction in spasticity and pressure sensitivity than those who will not receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* First-ever unilateral stroke;
* hemiplegia resulting from stroke;
* unilateral equinovarus gait with independent walk;
* able to ambulate without supporting devices.

Exclusion Criteria:

* recurrent stroke;
* previous treatment with nerve blocks, motor point injections with neurolytic agents for spasticity at any time, or with BTX-A in the previous 6 months
* not independent in the basic activities of daily living
* severe cognitive deficits;
* progressive or severe neurologic diseases;
* fear to needles;
* any contraindication for dry needling, e.g., anticoagulants, infections, bleeding, or psychotic.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Changes in spasticity before and after the intervention | Baseline and immediate after the inetrvention
  Spasticity in the affected ankle joint will be evaluated with the Modified Modified Ashworth Scale (MMAS). The examiner passively will move the ankle in dorsal-flexion direction, back and forth at least 5 times and will evaluate the degree of resistance to the movement on a scale from 0-4. This outcome will take 1 minute approximately.

SECONDARY OUTCOMES:
Changes in pressure pain sensitivity before and after the intervention | Baseline and immediate after the inetrvention
  Pressure pain sensitivity will be bilaterally assessed with a mechanical pressure algometer (Pain Diagnosis and Treatment Inc, New York, USA) over the deltoid muscle, the second metacarpal and the tibialis anterior muscle to determine changes in widespread pressure sensitivity. This outcome will take 5 minute approximately.
Changes in baropodometry outcomes before and after the intervention | Baseline and immediate after the inetrvention
  The following baropodometric data will be bilaterally collected from each patient: support surface (cm2), percentage of load (%) and force distribution (%) of both forefoot and rear foot. Additionally, we will also calculate mean and maximum pressure of each foot, affected and non-affected. This outcome will take 10 minutes approximately.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Salom, PT, MSc, Principal Investigator — Universidad Rey Juan Carlos; César Fernández-de-las-Peñas, PT, DO, PhD, Study Chair — Universidad Rey Juan Carlos
Locations (1):
- Universidad Rey Juan Carlos, Alcorcón, Madrid, Spain